CLINICAL TRIAL: NCT01119937
Title: A 52-week Treatment, Multi-center, Randomized, Open Label, Parallel Group Study to Assess the Long Term Safety and Tolerability of NVA237 (50µg o.d.) Using Tiotropium (18µg o.d.) as an Active Control in Japanese Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Long Term Safety and Tolerability of NVA237 Versus Tiotropium in Japanese Patients
Acronym: GLOW4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNVA237A1302
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; NVA237
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

ARMS (2):
- NVA237 (Experimental): 50µg once daily
  Interventions: Drug: NVA237
- Tiotropium (Experimental): 18µg once daily
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: NVA237 — 50µg capsules for inhalation, delivered via a single dose dry powder inhaler (Concept 1®)
  Arms: NVA237
Drug: Tiotropium — 18µg capsules for inhalation, delivered via HandiHaler®
  Arms: Tiotropium

SUMMARY:
This is a 52-week, multi-center, randomized, open label, parallel group study to assess the long term safety and tolerability of once-daily NVA237, using tiotropium as an active control, in Japanese patients with moderate to severe chronic obstructive pulmonary disease (COPD) .

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe stable COPD (Stage II or Stage III) according to the Gold Guideline 2008.
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* Patients with a post-bronchodilator FEV1 ≥30% and < 80% of the predicted normal, and postbronchodilator FEV1/FVC < 0.7 at Visit 2 (day -7)

Exclusion Criteria:

* Pregnant women or nursing mothers or women of child-bearing potential not using an acceptable method of contraception
* Patients requiring long term oxygen therapy
* Patients who have had a lower respiratory tract infection within 6 weeks prior to Visit 1
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions
* Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
* Patients in the active phase of a supervised pulmonary rehabilitation program
* Patients contraindicated for tiotropium or ipratropium treatment or who have shown an untoward reaction to inhaled anticholinergic agents
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (36):
- Japan (36):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Ōnojō, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Takarazuka, Hyōgo
  - Novartis Investigative Site, Yabu, Hyōgo
  - Novartis Investigative Site, Inashiki-gun, Ibaraki
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Sashima-gun, Ibaraki
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Uji, Kyoto
  - Novartis Investigative Site, Matsusaka, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Kasaoka, Okayama-ken
  - Novartis Investigative Site, Tsuyama, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Shimotsuka-gun, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Nakano-ku, Tokyo
  - Novartis Investigative Site, Ohta-ku, Tokyo
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Ube, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 211 participants entered screening. 163 participants entered treatment.
Period: Overall Study
Arm/Group | NVA237 | Tiotropium
Started | 123 | 40
Completed | 104 | 33
Not Completed | 19 | 7
Not completed — Adverse Event | 11 | 5
Not completed — Protocol deviation | 3 | 1
Not completed — Unsatisfactory therapeutic effect | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 | Tiotropium | Total
Number analyzed (Participants) | 123 | 40 | 163
Age Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.29) | 69.4 (7.48) | 68.7 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 121 | 38 | 159

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events or Death
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal lab finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgments of the investigators represent significant hazards.
Time Frame: 52 weeks
Population: Safety population - all patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
participants
  Adverse events | 102 | 33
  Serious adverse events | 16 | 6
  Death | 0 | 0

2. Secondary Outcome: Change in Pre-dose FEV1 From Baseline
Description: Pre-dose FEV1 is defined as the average of the measurements at 45 and 15 minutes pre-dose.
Time Frame: Weeks 12, 24, 36 and 52
Population: Intent-to-treat (ITT) population - included all randomized patients who received at least one dose of study drug. Only participants with measurements at both baseline and the specified timepoint were included in the analysis for the specific timepoint.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 110 | 37
liters
  Week 12 | 0.101 (0.1455) | 0.173 (0.1976)
  Week 24 | 0.094 (0.1614) | 0.144 (0.1435)
  Week 36 (n = 106, 36) | 0.084 (0.1558) | 0.112 (0.2200)
  Week 52 (n = 103, 33) | 0.068 (0.1829) | 0.127 (0.2566)

3. Secondary Outcome: Change in Pre-dose FVC From Baseline
Description: Pre-dose FVC is defined as the average of the measurements at 45 and 15 minutes pre-dose.
Time Frame: Weeks 12, 24, 36 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 110 | 37
liters
  Week 12 | 0.221 (0.3057) | 0.220 (0.3029)
  Week 24 | 0.218 (0.2798) | 0.179 (0.2285)
  Week 36 (n = 106, 36) | 0.208 (0.3204) | 0.146 (0.2547)
  Week 52 (n = 103, 33) | 0.195 (0.3739) | 0.126 (0.2889)

4. Secondary Outcome: Time From Randomization Until the Start of the First Moderate or Severe COPD Exacerbation
Description: Moderate COPD exacerbations were defined as: worsening of 2 or more of the following major symptoms for at least 2 consecutive days - dyspnea, sputum volume and sputum purulence; OR a worsening of any 1 major symptom with any 1 of the following minor symptoms for at least 2 consecutive days - sore throat, colds, fever without other cause, increased cough or increased wheeze, requiring treatment with systemic glucocorticosteroids or antibiotics or both. Severe COPD exacerbations were defined as: conditions for Moderate COPD exacerbation and hospitalization was required. Participants who withdraw from the study and do not experience a moderate or severe exacerbation are censored at the date of withdrawal. Participants who complete the study and do not experience a moderate or severe exacerbation are censored at the completion visit date.
Time Frame: 52 weeks
Population: Intent-to-treat (ITT) population - included all randomized patients who received at least one dose of study drug
Measure: Number; unit: days
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
days | 362 [2 to 372] | 359 [4 to 368]

5. Secondary Outcome: Number of Patients With Moderate or Severe COPD Exacerbations
Description: Moderate COPD exacerbations were defined as: worsening of 2 or more of the following major symptoms for at least 2 consecutive days - dyspnea, sputum volume and sputum purulence; OR a worsening of any 1 major symptom with any 1 of the following minor symptoms for at least 2 consecutive days - sore throat, colds, fever without other cause, increased cough or increased wheeze, requiring treatment with systemic glucocorticosteroids or antibiotics or both. Severe COPD exacerbations were defined as: conditions for Moderate COPD exacerbation and hospitalization was required.
Time Frame: 52 weeks
Population: Intent-to-treat (ITT) population - included all randomized patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
participants
  0 exacerbations | 99 | 31
  1 exacerbation | 17 | 5
  2 exacerbations | 5 | 3
  3 exacerbations | 1 | 0
  > = 4 exacerbations | 1 | 1

6. Secondary Outcome: Change in St. George Respiratory Questionnaire From Baseline
Description: SGRQ is a health related quality of life questionnaire consisting of 51 items in three components: symptoms, activity, and impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 121 | 40
score on a scale
  Week 12 | -2.57 (8.506) | -2.31 (13.654)
  Week 24 | -1.77 (9.466) | -3.24 (12.908)
  Week 36 | -2.54 (9.614) | -0.93 (14.214)
  Week 52 | -2.68 (10.505) | 0.36 (15.389)

7. Secondary Outcome: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication Over the Whole Treatment Period
Description: Patients recorded rescue medication use in a paper patient diary. If a patient required the use of salbutamol as rescue medication due to an increase in COPD symptoms, the number of inhalations (puffs) taken was recorded in the patient diary.
Time Frame: 52 weeks
Population: Intent-to-treat (ITT) population - included all randomized patients who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: change in puffs
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
change in puffs | -0.16 (1.039) | -0.27 (0.859)

8. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Hematology Values at Any Timepoint Over the Whole Treatment Period
Description: Clinically notable hematology values were: hemoglobin - male <11.5g/dL, female <9.5 g/dL; hematocrit - male <37%, female <32%; white cell count - <2800µL or >16000µL; platelets - <7.5 10*4/µL or >70.0 10*4/µL
Time Frame: 52 weeks
Population: Safety population - all patients who received at least one dose of study drug. Only participants with the required measurements were included for each specific value.
Measure: Number; unit: participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
participants
  Hemoglobin - male (n = 121, 38) | 3 | 2
  Hemoglobin - female (n = 121, 38) | 0 | 0
  Hematocrit - male (n = 121, 38) | 3 | 4
  Hematocrit - female (n = 121, 38) | 0 | 0
  White cell count - <2800/µL | 0 | 1
  White cell count - >16000/µL | 0 | 0
  Platelets - <7.5 10*4/µL | 1 | 0
  Platelets - >70.0 10*4/µL | 0 | 0

9. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Biochemistry Values at Any Timepoint Over the Whole Treatment Period
Description: Clinically notable biochemistry values were: total protein - <4.0 g/dL or >9.5 g/dL; albumin <2.5 g/dL; bilirubin (total) >1.9 mg/dL; BUN >27 mg/dL; creatinine >1.99 mg/dL; AST >3 x ULN U/L; ALT >3 x ULN U/L; ALP >3 x ULN U/L; y-GTP >3 x ULN U/L; sodium <125 mEq/L or >160 mEq/L; potassium <3.0 mEq/L or >6.0 mEq/L; glucose <51.0 mg/dL or >180.0 mg/dL
Time Frame: 52 weeks
Population: Safety population - all patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
participants
  Total protein - <4.0 g/dL | 0 | 0
  Total protein - >9.5 g/dL | 0 | 0
  Albumin - <2.5 g/dL | 0 | 0
  Bilirubin (total) - >1.9 mg/dL | 2 | 0
  BUN - >27 mg/dL | 3 | 0
  Creatinine - >1.99 mg/dL | 0 | 0
  AST - >3 x ULN U/L | 1 | 0
  ALT - >3 x ULN U/L | 0 | 0
  ALP - >3 x ULN U/L | 0 | 1
  Y-GTP - >3 x ULN U/L | 5 | 4
  Sodium - <125 mEq/L | 0 | 0
  Sodium - >160 mEq/L | 0 | 0
  Potassium - <3.0 mEq/L | 1 | 0
  Potassium - >6.0 mEq/L | 0 | 0
  Glucose - <51.0 mg/dL | 0 | 0
  Glucose - >180.0 mg/dL | 11 | 3

10. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Vital Signs Values at Any Timepoint Over the Whole Treatment Period
Description: Clinically notable vital sign values were: pulse rate - low, <40 bpm or <=50 bpm and decrease from baseline >=15bpm; pulse rate high, >130 bpm or >=120bpm and increase from baseline >=15 bpm. Systolic blood pressure - low, <75 mmHg or <=90 mmHg and decrease from baseline >=20 mmHg; high, >200 mmHg or >=180 mmHg and increase from baseline >=20 mmHg. Diastolic blood pressure - low, <40 mmHg or <=50 mmHg and decrease from baseline >=15 mmHg; high, >115 mmHg or >=105 mmHg and increase from baseline >=15 mmHg.
Time Frame: 52 weeks
Population: Safety population - all patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
participants
  Pulse rate - low | 0 | 1
  Pulse rate - high | 0 | 0
  Pulse rate - low or high | 0 | 1
  Systolic blood pressure - low | 0 | 0
  Systolic blood pressure - high | 1 | 0
  Systolic blood pressure - low or high | 1 | 0
  Diastolic blood pressure - low | 1 | 0
  Diastolic blood pressure - high | 2 | 0
  Diastolic blood pressure - low or high | 3 | 0

11. Secondary Outcome: Number of Patients With Notable Change From Baseline in Fridericia's QTc Values at Any Timepoint Over the Whole Treatment Period
Description: Clinically notable change from baseline was and increase from baseline of 30 or greater milliseconds (ms).
Time Frame: 52 weeks
Population: Safety population - all patients who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 123 | 40
participants
  Increase from baseline 30 to 60 ms | 6 | 1
  Increase from baseline >60 ms | 2 | 0

ADVERSE EVENTS:
Arm/Group | NVA237 | Tiotropium
Serious Adverse Events (participants affected / at risk) | 16/123 | 6/40
Other Adverse Events (participants affected / at risk) | 83/123 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=123) | Tiotropium (N=40)
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=123) | Tiotropium (N=40)
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 2
Cataract (Eye disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2
Gastric xanthoma (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 3
Gastritis atrophic (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Metaplasia (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 6 | 5
Eczema impetiginous (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Helicobacter infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 37 | 13
Oral herpes (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 6 | 1
Pneumonia (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1
Skin candida (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Upper respiratory tract infection bacterial (Infections and infestations) | 6 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Platelet count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 1
Dysuria (Renal and urinary disorders) | 3 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.